CLINICAL TRIAL: NCT03253614
Title: Auditive and Renal Long Term Outcomes - Risk After Aminoglycoside Therapy in Neonates (AURORA-study)
Brief Title: Auditive and Renal Long Term Outcomes - Risk After Aminoglycoside Therapy in Neonates (AURORA)
Acronym: AURORA
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Claus Klingenberg, Professor, University Hospital of North Norway
Other Study IDs: REK Nord 2016/1786
Record Dates: First submitted 2017-08-14; First posted 2017-08-18 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Hearing Loss; Gentamicin Adverse Reaction; Renal Tubular Disorder
MeSH Terms: conditions — Hearing Loss | interventions — Audiometry; Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine biomarkers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: 250 children aged 6-15 years exposed to gentamicin in the neonatal period
  Interventions: Diagnostic Test: Audiometry; Diagnostic Test: Urine biomarkers for renal tubular function; Diagnostic Test: Blood pressure
- Control group: 25 healthy children aged 6-15 years NOT exposed to gentamicin in the neonatal period
  Interventions: Diagnostic Test: Audiometry

INTERVENTIONS:
Diagnostic Test: Audiometry — Extended high-frequency (EHF; 9-16 kHz) audiometry
Diagnostic Test: Urine biomarkers for renal tubular function — Kidney Injury Molecule-1
  Groups: Exposed group
Diagnostic Test: Blood pressure — Blood pressure right arm, measured With standard Methods 3 times
  Groups: Exposed group

SUMMARY:
Gentamicin, in combination with a beta-lactam antibiotic, is commonly used for treatment of neonatal sepsis. Neonates have a high volume of distribution. It is a paradox that most neonatal dosing schedules still recommend lower gentamicin doses (4-5 mg/kg) than in older children (≥ 7 mg/kg). In the neonatal unit in Tromsø a simplified gentamicin high-dose (6 mg/kg) regimen has been in use since 2004.

The investigators have previously shown that this regimen was associated with low number of elevated trough levels, low numbers of prescription errors and no evidence for ototoxicity in the immediate neonatal period. However, the long-term safety of gentamicin therapy in neonates is not well studied when it comes to ototoxicity and possible nephrotoxicity.

The objective of the current study is therefore to perform a detailed hearing evaluation, including an extended high-frequency (EHF; 9-16 kHz) audiometry, in a follow-up study of children (participants) aged 6-15 years who were exposed to a high-dose gentamicin regimen in the neonatal period. Moreover, we will investigate blood pressure and urine biomarkers to assess renal tubular function. The aim is to include 250 children exposed to gentamicin in the neonatal period and a control group of 25 healthy children.

EHF audiometry is a more sensitive method for detecting ototoxic damage and provides evidence of ototoxicity before any hearing loss is detected by conventional systems. This is the background for choice of method.

The primary outcome is the difference in average hearing threshold in the EHF range between the control group and the exposed group.

Secondary outcomes are i) difference in average hearing threshold in the EHF range between the children with gentamicin trough levels > 1.0 mg/L versus those who had lower trough levels, ii) markers of renal tubular function (kidney injury molecule 1) and iii) blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Exposed to gentamicin therapy in the neonatal period and treated at neonatal unit at the University Hospital of North Norway

Exclusion Criteria:

* Not able to cooperate during an audiometry

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 6-15 years and Exposed to gentamicin therapy in the neonatal period and treated at neonatal unit at the University Hospital of North Norway.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Hearing threshold in the extended high-frequency range | Baseline
  kHz

SECONDARY OUTCOMES:
Urine biomarkers | Baseline
  Kidney injury molecule-1
Blood pressure right arm | Baseline
  mm Hg
Hearing threshold in the normal frequency range | Baseline
  kHz

CONTACTS AND LOCATIONS:
Overall Officials: Claus Klingenberg, MD, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available after publication of the first scientific report. Sharing of data will be done after a signed agreement.

REFERENCES:
- [Background] Fjalstad JW, Laukli E, van den Anker JN, Klingenberg C. High-dose gentamicin in newborn infants: is it safe? Eur J Pediatr. 2013 Nov 14. doi: 10.1007/s00431-013-2194-1. Online ahead of print. PMID 24233331
- [Background] Setiabudy R, Suwento R, Rundjan L, Yasin FH, Louisa M, Dwijayanti A, Simanjuntak E. Lack of a relationship between the serum concentration of aminoglycosides and ototoxicity in neonates. Int J Clin Pharmacol Ther. 2013 May;51(5):401-6. doi: 10.5414/CP201833. PMID 23557866
- [Derived] Rypdal V, Jorandli S, Hemmingsen D, Solbu MD, Klingenberg C. Exposure to an Extended-Interval, High-Dose Gentamicin Regimen in the Neonatal Period Is Not Associated With Long-Term Nephrotoxicity. Front Pediatr. 2021 Nov 30;9:779827. doi: 10.3389/fped.2021.779827. eCollection 2021. PMID 34917565
- [Derived] Hemmingsen D, Stenklev NC, Klingenberg C. Extended high frequency audiometry thresholds in healthy school children. Int J Pediatr Otorhinolaryngol. 2021 May;144:110686. doi: 10.1016/j.ijporl.2021.110686. Epub 2021 Mar 23. PMID 33838463
- [Derived] Hemmingsen D, Mikalsen C, Hansen AR, Fjalstad JW, Stenklev NC, Klingenberg C. Hearing in Schoolchildren After Neonatal Exposure to a High-Dose Gentamicin Regimen. Pediatrics. 2020 Feb;145(2):e20192373. doi: 10.1542/peds.2019-2373. Epub 2020 Jan 8. PMID 31915192